CLINICAL TRIAL: NCT02932410
Title: A Multicenter, Open-label, Randomized, Study With Single-arm Extension Period to Assess the Pharmacokinetics, Safety and Efficacy of Macitentan Versus Standard of Care in Children With Pulmonary Arterial Hypertension
Brief Title: A Study to Assess Whether Macitentan Delays Disease Progression in Children With Pulmonary Arterial Hypertension (PAH)
Acronym: TOMORROW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-055-312
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Results first posted 2025-09-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Macitentan (Experimental): Macitentan is administered once daily via oral route. Children less than (<) 2 years old (y.o.) will be assigned as a cohort to the macitentan group without randomization. The dose will be adjusted to the participant's age (for those < 2 y.o.) or to the participant's body weight (for those greater than or equal to (>=) 2 y.o.). single-arm extension period (SAEP) will start at end of core period (EOCP) visit and ends at end of study (EOS) visit.
  Interventions: Drug: Macitentan
- Standard-of-care (Other): Standard-of-care as per site's clinical practice which may comprise treatment with pulmonary arterial hypertension (PAH) non-specific treatment and/or up to two PAH-specific medications excluding macitentan and intravenous/subcutaneous (IV/SC) prostanoids.
  Interventions: Other: Standard-of-care

INTERVENTIONS:
Drug: Macitentan — Dispersible tablet; Oral use
  Other Names: ACT-064992
  Arms: Macitentan
Other: Standard-of-care — Standard-of-care as per site's clinical practice which may comprise treatment with PAH non-specific treatment and/or up to two PAH-specific medications excluding macitentan and IV/SC prostanoids.
  Arms: Standard-of-care

SUMMARY:
This is a prospective, multicenter, open-label, randomized, controlled, parallel Phase 3 study with an open-label single-arm extension period to evaluate pharmacokinetics (PK), safety and efficacy of macitentan in children with pulmonary arterial hypertension (PAH).

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent by the parent(s) or legally designated representative and assent from developmentally capable children prior to initiation of any study-mandated procedure
* Males or females between greater than or equal to (>=) 1 month and less than (<) 18 years of age
* Participants with body weight >= 3.5 kilograms (kg) at randomization
* Pulmonary arterial hypertension (PAH) diagnosis confirmed by historical RHC (mPAP greater than or equal to [>=] 25 millimeters of mercury [mmHg], and Pulmonary artery wedge pressure [PAWP] less than or equal to [<=] 15 mmHg, and Pulmonary vascular resistance index [PVRi] greater than [>] 3 WU × m2), where in the absence of pulmonary vein obstruction and/or significant lung disease PAWP can be replaced by Left atrium pressure [LAP] or Left ventricular end diastolic pressure [LVEDP] (in absence of mitral stenosis) assessed by heart catheterization
* PAH belonging to the Nice 2013 Updated Classification Group 1 (including participants with Down Syndrome) and of following etiologies: idiopathic PAH; heritable PAH; PAH associated with congenital heart disease (CHD); Drug or toxin induced PAH; PAH associated with HIV; PAH associated with connective tissue diseases (PAH-aCTD); and World health organization (WHO) Functional class I to III
* Females of childbearing potential must have a negative pregnancy test at Screening and at Baseline, and must agree to undertake monthly pregnancy tests, and to use a reliable method of contraception (if sexually active) up to the end of study (EOS)

Key Exclusion Criteria:

* Participants with PAH due to portal hypertension, schistosomiasis, or with pulmonary veno-occlusive disease and/or pulmonary capillary hemangiomatosis, and persistent pulmonary hypertension of the newborn
* Participants with PAH associated with Eisenmenger syndrome, or with moderate to large left-to-right shunts
* Participants receiving a combination of > 2 PAH-specific treatments at randomization.
* Treatment with intravenous (IV) or subcutaneous (SC) prostanoids within 4 weeks before randomization, unless given for vasoreactivity testing
* Hemoglobin or hematocrit <75 percent (%) of the lower limit of normal range
* Serum Aspartate aminotransferase (AST) and/or Alanine aminotransferase (ALT) greater than (>) 3 times the upper limit of normal range
* Pregnancy (including family planning) or breastfeeding.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol
* Severe hepatic impairment, for example Child-Pugh Class C
* Clinical signs of hypotension which in the investigator's judgment would preclude initiation of a PAH-specific therapy
* Severe renal insufficiency (estimated creatinine clearance <30 mL/min or serum creatinine >221 micro-moles per liter [micro-mol/L])
* Participants with known diagnosis of bronchopulmonary dysplasia

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2025-11-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (85):
- United States (20):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - UCLA Children's Heart Center, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Riley Hospital For Children, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Detroit Medical Center, Detroit, Michigan
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Children's Heart Center, Las Vegas, Nevada
  - Columbia University Medical Center - PIN, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Childrens Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Royal Children's Hospital Melbourne - PIN, Parkville
  - Lady Cilento Children's Hospital, South Brisbane
  - Children's Hospital at Westmead, Westmead
- Austria (3):
  - Medizinische Universität Graz, Graz
  - Landes Frauen Und Kinderklinik Linz, Linz
  - Medizinische Universitat Wien, Linz
- Irmandade Da Santa Casa de Misericórdia de São Paulo, São Paulo, Brazil
- Sainte Justine Hospital, Montreal, Canada
- China (4):
  - Beijing Anzhen Hospital of The Capital University of Medical Sciences, Beijing
  - Qingdao Women and Children's Hospital, Qingdao
  - Childrens Hospital of Shanghai, Shanghai
  - Shanghai Children's Medical Center, Shanghai
- Colombia (2):
  - Fundacion Santa Fe de Bogota, Bogotá
  - Centro Medico Imbanaco de Cali SA, Cali
- HUS Uusi lastensairaala, Helsinki, Finland
- France (4):
  - Hôpital de la Timone Enfants, Marseille
  - Groupe Hospitalier Necker Enfants Malades, Paris
  - Hôpital Haut-Lévêque - Hôpital cardiologique, Pessac
  - Hôpital Des Enfants, Toulouse
- Gottsegen Gyorgy Orszagos Kardiologiai Intezet, Budapest, Hungary
- Israel (3):
  - Rambam Medical Center - PPDS, Haifa
  - Schneider Children's Medical Center of Israel - PIN, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Malaysia (2):
  - Institut Jantung Negara, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- Mexico (5):
  - CICUM San Miguel, Guadalajara
  - Instituto Nacional de Pediatría, Mexico City
  - Instituto Nacional de Cardiologia Dr. Ignacio Chavez, Mexico City
  - Operadora de Hospitales Angeles SA de CV Hospital Angeles Lomas, México
  - Unidad de Investigación Clínica En Medicina SC, Monterrey
- Philippines (2):
  - Makati Medical Center, Makati City
  - Philippine Heart Center, Quezon City
- Poland (3):
  - Szpital Kliniczny im. Karola Jonschera Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Instytut Pomnik - Centrum Zdrowia Dziecka, Warsaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu Osrodek Badawczo-Rozwojowy, Wroclaw
- Portugal (4):
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital de Santa Cruz, Carnaxide
  - Centro Hospitalar E Universitário de Coimbra EPE, Coimbra
  - Hospital Santa Marta, Lisbon
  - Centro Hospitalar de Sao Joao EPE, Porto
- Russia (7):
  - Research Institute of Complex Cardiovascular Pathology, Kemerovo
  - GBUZ Children's Hospital named after Bashlyaeva Z.A. Moscow, Moscow
  - Russian National Research Medical University n.a. N.I.Pirogov, Moscow
  - Novosibirsk Research Institue of Blood Circulation Pathology n.a. E.N. Meshalkin, Novosibirsk
  - Saint Petersburg State Pediatric Medical Academy, Saint Petersburg
  - Clinical Hospital №1, Tyumen
  - Bashkiria State Medical University, Ufa
- South Africa (2):
  - University of The Free State, Bloemfontein
  - Inkosi Albert Luthuli Central Hospital, Durban
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
- Spain (7):
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - C.H. Regional Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Maharaj Nakorn Chiang Mai Chiang Mai University, Chiang Mai, Thailand
- Ukraine (3):
  - MI Dnipropetrovsk Specialized Clin. Med. Center of Mother and Child n.a. prof. M.F. Rudnev of DRC, Dnipro
  - Municipal Institution of Health Care Regional Children's Clinical Hospital, Kharkiv
  - MI Scientific Practical Medical Center for Children Cardiology and Cardiosurgery of MOH of Ukraine, Kyiv
- Vietnam (4):
  - Hanoi Heart Hospital, Hanoi
  - Hanoi Medical University Hospital, Hanoi
  - Children's Hospital 1, Ho Chi Minh City
  - Tam Duc Hospital, Ho Chi Minh City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants up to less than (<) 18 years at the time of enrolment were classified into one of the treatment arms: Macitentan (greater than or equal to [>=] 2 years), standard of care (SOC: >=2 years), Macitentan (<2 years) or China Single Arm Cohort (>=12 years).
Pre-assignment Details: Participants from 2 to <18 years were randomized (1:1) to either macitentan or to SoC. Randomization was stratified by ongoing/planned Endothelin Receptor Antagonist treatment at randomization (yes vs no) and by WHO Functional Class (FC) at randomization (FC I/II vs FC III). Participants <2 years or participants in China single arm cohort were assigned to macitentan arm without randomization. Adverse events are reported until end of core period analysis which is beyond primary completion date.
Groups:
- Macitentan (JNJ-67896062) (>=2 Years): Randomized participants aged >=2 years received macitentan orally (dispersible tablet reconstituted in water) once daily based on their body weight (BW): 3.5 milligrams (mg) for BW >=10 kilograms (kg) and <15 kg, 5.0 mg for >=15 kg and <25 kg, 7.5 mg for >=25 kg and <50 kg, and 10.0 mg for >=50 kg. Every 12 weeks body weight was checked for potential dose adjustment. Phosphodiesterase Type 5 inhibitor (PDE-5i) was the only allowed PAH-specific background medication until disease progression. Participants received treatment from Day 1 up to 312.4 weeks.
- Standard of Care (SoC; >=2 Years): Randomized participants aged >=2 years continued their SoC as per site's clinical practice which comprised treatment with the pulmonary arterial hypertension (PAH) non-specific treatment and/or up to 2 PAH-specific medications excluding macitentan and intravenous (IV)/subcutaneous (SC) prostanoids. Participants continued to receive the PDE-5i (sildenafil and tadalafil), or other PAH-specific treatment such as an ERA (bosentan and ambrisentan) or oral prostanoids (soluble guanylate cyclase stimulators [riociguat]), which was ongoing at the time of randomization. Additional PAH-specific therapy other than macitentan and IV or SC prostanoids initiated prior to randomization was continued. Participants received treatment from Day 1 up to 316.4 weeks. For participants with disease progression, crossover to macitentan was offered after confirmation of a disease progression event by the blinded Clinical Event Committee.
- Macitentan (JNJ-67896062) (<2 Years): Enrolled participants aged <2 years received macitentan 2.5 mg once daily orally (dispersible tablet reconstituted in water). Oral or inhaled prostanoid treatment were allowed as PAH-specific background therapy. Participants received treatment from Day 1 up to 72.9 weeks.
- China Single-arm Cohort (>=12 to <18 Years): Enrolled participants aged >=12 to <18 years received macitentan orally (dispersible tablet reconstituted in water) once daily based on their body weight (BW): 3.5 milligrams (mg) for BW >=10 kilograms (kg) and <15 kg, 5.0 mg for >=15 kg and <25 kg, 7.5 mg for >=25 kg and <50 kg and 10.0 mg for >=50 kg. Every 12 weeks body weight was checked for potential dose adjustment. Phosphodiesterase Type 5 (PDE-5) inhibitor was the only allowed PAH-specific background medication until disease progression. Participants received treatment from Day 1 up to 48.29 weeks.
Period: Overall Study
Arm/Group | Macitentan (JNJ-67896062) (>=2 Years) | Standard of Care (SoC; >=2 Years) | Macitentan (JNJ-67896062) (<2 Years) | China Single-arm Cohort (>=12 to <18 Years)
Started | 73 | 75 | 9 | 8
Treated | 72 | 75 | 9 | 8
Crossed Over to Macitentan Treatment | 0 | 8 | 0 | 0
Completed | 59 | 60 | 8 | 8
Not Completed | 14 | 15 | 1 | 0
Not completed — Death | 7 | 6 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Parent/Subjects decision | 6 | 6 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Macitentan (JNJ-67896062) (>=2 Years) | Standard of Care (SoC; >=2 Years) | Macitentan (JNJ-67896062) (<2 Years) | China Single-arm Cohort (>=12 to <18 Years) | Total
Number analyzed (Participants) | 73 | 75 | 9 | 8 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (4.43) | 9 (4.32) | 1.7 (0.27) | 12.9 (1.13) | 9.4 (4.65)
Age, Customized [Count of Participants; unit: Participants]
  >= 0 to < 0.5 years | 0 | 0 | 0 | 0 | 0
  >= 0.5 to < 2 years | 0 | 0 | 9 | 0 | 9
  >= 2 to < 6 years | 13 | 22 | 0 | 0 | 35
  >= 6 to < 12 years | 29 | 32 | 0 | 0 | 61
  >= 12 to < 18 years | 31 | 21 | 0 | 8 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 38 | 1 | 4 | 93
  Male | 23 | 37 | 8 | 4 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 22 | 2 | 0 | 48
  Not Hispanic or Latino | 47 | 51 | 6 | 8 | 112
  Unknown or Not Reported | 2 | 2 | 1 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 15 | 22 | 3 | 8 | 48
  Black or African American | 1 | 1 | 2 | 0 | 4
  White | 44 | 32 | 2 | 0 | 78
  Unknown or Not Reported | 1 | 2 | 0 | 0 | 3
  Other | 12 | 18 | 2 | 0 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 2 | 2 | 0 | 0 | 4
  BRAZIL | 1 | 1 | 0 | 0 | 2
  CHINA | 1 | 0 | 0 | 8 | 9
  COLOMBIA | 7 | 7 | 0 | 0 | 14
  FRANCE | 1 | 2 | 0 | 0 | 3
  HUNGARY | 3 | 1 | 1 | 0 | 5
  ISRAEL | 1 | 2 | 0 | 0 | 3
  MALAYSIA | 0 | 0 | 1 | 0 | 1
  MEXICO | 15 | 14 | 2 | 0 | 31
  PHILIPPINES | 3 | 4 | 2 | 0 | 9
  POLAND | 2 | 2 | 0 | 0 | 4
  PORTUGAL | 3 | 1 | 1 | 0 | 5
  RUSSIAN FEDERATION | 7 | 6 | 0 | 0 | 13
  Korea, Republic of | 4 | 3 | 0 | 0 | 7
  SPAIN | 3 | 2 | 0 | 0 | 5
  THAILAND | 2 | 2 | 0 | 0 | 4
  UKRAINE | 8 | 7 | 0 | 0 | 15
  UNITED STATES | 6 | 6 | 2 | 0 | 14
  VIETNAM | 4 | 13 | 0 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Participants >=2 Years of Age: Observed Steady-State Trough (Pre-dose) Plasma Concentration of Macitentan and Aprocitentan (Active Metabolite) at Week 12 Based on Body Weight
Description: Observed steady-state trough (pre-dose) plasma concentration of macitentan and aprocitentan (active metabolite) at Week 12 based on body weight were reported. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Pre-dose at Week 12
Population: The Pharmacokinetics (PK) 1 set included all participants aged >=2 years randomized to and treated with macitentan, for whom a PK blood sample at trough had been taken and who did not deviate from the protocol in a way that affected the evaluation of the PK trough endpoints. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure and "n"(number analyzed) signifies number of participants analyzed for specified categories.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Macitentan (JNJ-67896062) (>=2 Years)
Number analyzed (Participants) | 47
nanograms per milliliter (ng/mL)
  Macitentan: >=10 kg and <15 kg: number analyzed (Participants) | 6
  Macitentan: >=10 kg and <15 kg | 150.133 (67.5742)
  Macitentan: >=15 kg and <25 kg: number analyzed (Participants) | 12
  Macitentan: >=15 kg and <25 kg | 153.892 (108.3185)
  Macitentan: >=25 kg and <50 kg: number analyzed (Participants) | 14
  Macitentan: >=25 kg and <50 kg | 200.975 (151.6511)
  Macitentan: >=50 kg: number analyzed (Participants) | 15
  Macitentan: >=50 kg | 208.067 (92.4246)
  Aprocitentan: >=10 kg to <15 kg: number analyzed (Participants) | 6
  Aprocitentan: >=10 kg to <15 kg | 1165.000 (390.7628)
  Aprocitentan: >=15 kg and <25 kg: number analyzed (Participants) | 12
  Aprocitentan: >=15 kg and <25 kg | 859.333 (217.2926)
  Aprocitentan: >=25 kg and <50 kg: number analyzed (Participants) | 14
  Aprocitentan: >=25 kg and <50 kg | 980.857 (391.3308)
  Aprocitentan: >=50 kg: number analyzed (Participants) | 15
  Aprocitentan: >=50 kg | 1011.267 (288.3632)

2. Primary Outcome: Participants >=2 Years of Age: Observed Steady-State Trough (Pre-dose) Plasma Concentration of Macitentan and Aprocitentan (Active Metabolite) at Week 12 Based on Age Group
Description: Observed steady-state trough (pre-dose) plasma concentration of macitentan and aprocitentan (active metabolite) at Week 12 based on age group were reported. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Pre-dose at Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Macitentan (JNJ-67896062) (>=2 Years)
Number analyzed (Participants) | 47
nanograms per milliliter (ng/mL)
  Macitentan: >=2 to <6 years: number analyzed (Participants) | 9
  Macitentan: >=2 to <6 years | 159.767 (84.5424)
  Macitentan: >=6 to <12 years: number analyzed (Participants) | 19
  Macitentan: >=6 to <12 years | 184.792 (148.2530)
  Macitentan: >=12 to <18 years: number analyzed (Participants) | 19
  Macitentan: >=12 to <18 years | 196.484 (88.1549)
  Aprocitentan: >=2 to <6 years: number analyzed (Participants) | 9
  Aprocitentan: >=2 to <6 years | 1063.333 (376.4173)
  Aprocitentan: >=6 to <12 years: number analyzed (Participants) | 19
  Aprocitentan: >=6 to <12 years | 957.211 (335.0858)
  Aprocitentan: >=12 to <18 years: number analyzed (Participants) | 19
  Aprocitentan: >=12 to <18 years | 970.842 (298.5151)

3. Primary Outcome: Participants <2 Years of Age: Observed Steady-State Trough (Pre-dose) Plasma Concentration of Macitentan and Aprocitentan (Active Metabolite) at Week 4
Description: Observed steady-state trough (pre-dose) plasma concentration of macitentan and aprocitentan (active metabolite) at Week 4 were reported. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Pre-dose at Week 4
Population: PK Set 3 included all participants aged <2 years and treated with macitentan for whom a PK blood sample had been taken and who did not deviate from the protocol in a way that might affect the evaluation of the PK endpoints.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Macitentan (JNJ-67896062) (<2 Years)
Number analyzed (Participants) | 9
ng/mL
  Macitentan | 101.822 (91.9652)
  Aprocitentan | 707.089 (465.5760)

4. Primary Outcome: Participants From China With >=12 to <18 Years of Age: Observed Steady-State Trough (Pre-dose) Plasma Concentration of Macitentan and Aprocitentan (Active Metabolite) at Week 12
Description: Observed steady-state trough (pre-dose) plasma concentration of macitentan and aprocitentan (active metabolite) at Week 12 were reported.
Time Frame: Pre-dose at Week 12
Population: PK Analysis Set China (PK CHN) included all participants >=12 years to <18 years who were treated with macitentan, for whom a PK blood sample has been taken and who did not deviate from the protocol in a way that might affect the evaluation of the PK endpoints.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | China Single-arm Cohort (>=12 to <18 Years)
Number analyzed (Participants) | 8
ng/mL
  Macitentan | 201.61 (116.685)
  Aprocitentan | 1313.75 (293.644)

5. Secondary Outcome: Time to the First Clinical Event Committee (CEC)-Confirmed Disease Progression Event
Time Frame: Baseline (Day 1) up to end of core study period (EOCP; up to 7.08 years)
Reporting Status: Not Posted, anticipated posting 2026-11

6. Secondary Outcome: Time to First CEC-confirmed Hospitalization for PAH
Time Frame: Baseline (Day 1) up to EOCP (up to 7.08 years)
Reporting Status: Not Posted, anticipated posting 2026-11

7. Secondary Outcome: Time to CEC-confirmed Death Due to PAH
Time Frame: Baseline (Day 1) up to EOCP (up to 7.08 years)
Reporting Status: Not Posted, anticipated posting 2026-11

8. Secondary Outcome: Time to Death (All Causes)
Time Frame: Baseline (Day 1) up to 7.26 years
Reporting Status: Not Posted, anticipated posting 2026-11

9. Secondary Outcome: Percentage of Participants With World Health Organization (WHO) Functional Class (FC) I or II Versus III or IV
Time Frame: At Weeks 12 and 24
Reporting Status: Not Posted, anticipated posting 2026-11

10. Secondary Outcome: Change From Baseline in N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) at Weeks 12 and 24
Time Frame: Baseline (Day 1), Weeks 12 and 24
Reporting Status: Not Posted, anticipated posting 2026-11

11. Secondary Outcome: Change From Baseline in Mean Daily Time Spent in Moderate to Vigorous Physical Activity as Measured by Accelerometry at Week 48
Time Frame: Baseline (Day 1), Week 48
Reporting Status: Not Posted, anticipated posting 2026-11

12. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) Normalized Tricuspid Annular Plane Systolic Excursion (TAPSE) Measured by Echocardiography at Week 24
Time Frame: Baseline (Day 1), Week 24
Reporting Status: Not Posted, anticipated posting 2026-11

13. Secondary Outcome: Change From Baseline in Left Ventricular Eccentricity Index (LVEI) Measured by Echocardiography at Week 24
Time Frame: Baseline (Day 1), Week 24
Reporting Status: Not Posted, anticipated posting 2026-11

14. Secondary Outcome: Change From Baseline in Quality of Life Measured by Pediatric Quality of Life Inventory Version 4.0 (PedsQL 4.0) Generic Core Scales Short Form (SF-15)
Time Frame: Baseline (Day 1), Week 24
Reporting Status: Not Posted, anticipated posting 2026-11

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline (Day 1) up to 7.26 years
Reporting Status: Not Posted, anticipated posting 2026-11

16. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Time Frame: Baseline (Day 1) up to 7.26 years
Reporting Status: Not Posted, anticipated posting 2026-11

17. Secondary Outcome: Number of Participants With AEs Leading to Premature Discontinuation of Macitentan or Standard of Care (SoC)
Time Frame: Baseline (Day 1) up to 7.26 years
Reporting Status: Not Posted, anticipated posting 2026-11

18. Secondary Outcome: Number of Participants With AEs of Special Interest
Time Frame: Baseline (Day 1) up to 7.26 years
Reporting Status: Not Posted, anticipated posting 2026-11

19. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Time Frame: Baseline (Day 1) up to 7.26 years
Reporting Status: Not Posted, anticipated posting 2026-11

20. Secondary Outcome: Change From Baseline in Selected Laboratory Parameters
Time Frame: Baseline (Day 1) up to 7.26 years
Reporting Status: Not Posted, anticipated posting 2026-11

21. Secondary Outcome: Change From Baseline in Vital Signs (Blood Pressure, Heart Rate)
Time Frame: Baseline (Day 1) up to 7.26 years
Reporting Status: Not Posted, anticipated posting 2026-11

22. Secondary Outcome: Change From Baseline in Growth Variable
Time Frame: Baseline (Day 1) up to 7.26 years
Reporting Status: Not Posted, anticipated posting 2026-11

23. Secondary Outcome: Change From Baseline in Sexual Maturation Measured by Tanner Stage
Time Frame: Baseline (Day 1) up to 7.26 years
Reporting Status: Not Posted, anticipated posting 2026-11

ADVERSE EVENTS:
Time Frame: All cause mortality: From screening (-6 weeks) up to 7.26 years; SAEs and Non-SAEs: Baseline (Day 1) up to end of core study period (EOCP; up to 7.08 years)
Description: All-cause mortality: FAS3 participants (FAS1 + FAS2) + FAS CHN participants (aged >= 12 years, assigned to macitentan without randomization). SAEs and other AEs: SAS3 (SAS1 + SAS2) + Safety CHN participants (aged >= 12 years, received at least 1 dose of macitentan)
Groups:
- Macitentan (JNJ67896062) (<2 Years): Enrolled participants aged <2 years received macitentan 2.5 mg once daily orally (dispersible tablet reconstituted in water). Oral or inhaled prostanoid treatment were allowed as PAH-specific background therapy. Participants received treatment from Day 1 up to 72.9 weeks.
- SOC (>=2 Years) Crossover to Macitentan: Participants aged >=2 years randomized to SoC arm and who had Clinical Event Committee-confirmed disease progression were offered to cross-over to macintentan treatment by signing a separate informed consent, if they agreed per investigator judgment. Eligible participants received macitentan orally (dispersible tablet reconstituted in water) once daily based on their BW: 3.5 mg for BW >=10 kg and <15 kg, 5.0 mg for >=15 kg and <25 kg, 7.5 mg for >=25 kg and <50 kg and 10.0 mg for >=50 kg. Every 12 weeks body weight was checked for potential dose adjustment. Participants received treatment from Day of disease confirmation up to 107 weeks.
Arm/Group | Macitentan (JNJ-67896062) (>=2 Years) | Macitentan (JNJ67896062) (<2 Years) | Standard of Care (SoC; >=2 Years) | SOC (>=2 Years) Crossover to Macitentan | China Single-arm Cohort (>=12 to <18 Years)
All-Cause Mortality (participants affected / at risk) | 7/73 | 0/9 | 6/75 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 26/72 | 4/9 | 21/75 | 0/8 | 1/8
Other Adverse Events (participants affected / at risk) | 60/72 | 6/9 | 44/75 | 5/8 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan (JNJ-67896062) (>=2 Years) (N=72) | Macitentan (JNJ67896062) (<2 Years) (N=9) | Standard of Care (SoC; >=2 Years) (N=75) | SOC (>=2 Years) Crossover to Macitentan (N=8) | China Single-arm Cohort (>=12 to <18 Years) (N=8)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0
Antiphospholipid Syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Cardiogenic Shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Right Ventricular Failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial Septal Defect (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Dengue Fever (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Febrile Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Mediastinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 2 | 1 | 0 | 0
Pneumonia Mycoplasmal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Salmonella Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Salpingo-Oophoritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 1 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Camptodactyly Acquired (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Systemic Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Brain Oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Status Epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urethral Stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Laryngeal Stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Systemic Sclerosis Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Extremity Necrosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan (JNJ-67896062) (>=2 Years) (N=72) | Macitentan (JNJ67896062) (<2 Years) (N=9) | Standard of Care (SoC; >=2 Years) (N=75) | SOC (>=2 Years) Crossover to Macitentan (N=8) | China Single-arm Cohort (>=12 to <18 Years) (N=8)
Anaemia (Blood and lymphatic system disorders) | 6 | 0 | 3 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 4 | 0 | 6 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 6 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0 | 8 | 0 | 0
Fatigue (General disorders) | 5 | 0 | 0 | 0 | 0
Feeling Abnormal (General disorders) | 0 | 0 | 1 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 4 | 0 | 4 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 7 | 1 | 3 | 1 | 0
Bronchitis (Infections and infestations) | 5 | 0 | 8 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Conjunctivitis (Infections and infestations) | 2 | 1 | 2 | 0 | 0
Covid-19 (Infections and infestations) | 11 | 2 | 6 | 1 | 0
Gastroenteritis (Infections and infestations) | 9 | 2 | 1 | 0 | 0
Influenza (Infections and infestations) | 8 | 0 | 4 | 0 | 1
Nasopharyngitis (Infections and infestations) | 14 | 0 | 12 | 1 | 0
Otitis Media Acute (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 5 | 0 | 6 | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 2 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 4 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 6 | 0 | 3 | 0 | 1
Suspected Covid-19 (Infections and infestations) | 1 | 0 | 2 | 1 | 0
Tonsillitis (Infections and infestations) | 4 | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 22 | 4 | 13 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 3 | 0 | 3 | 1 | 0
Varicella (Infections and infestations) | 2 | 0 | 1 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 | 1 | 3 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0
Anticoagulation Drug Level Increased (Investigations) | 0 | 0 | 1 | 1 | 0
Haemoglobin Decreased (Investigations) | 4 | 0 | 0 | 0 | 0
N-Terminal Prohormone Brain Natriuretic Peptide Increased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight Increased (Investigations) | 2 | 0 | 0 | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 6 | 0 | 2 | 1 | 0
Headache (Nervous system disorders) | 14 | 0 | 9 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 5 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 9 | 2 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 4 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the Sponsor for review at least 60 days before submission for publication or presentation. If requested by the Sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT02932410/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT02932410/SAP_001.pdf